CLINICAL TRIAL: NCT00834327
Title: A Randomized, Double-Blind, Placebo-Controlled Four Week Study of the Efficacy and Safety of Four Doses (0.05 mg, 0.1 mg, 0.25 mg, 0.5 mg) of Aplindore MR Tablets vs. Placebo in Idiopathic Restless Legs Syndrome.
Brief Title: Efficacy and Safety Study of Aplindore in Patients With Restless Legs Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Neurogen acquired by Ligand Pharmaceuticals - no further support for the study. No safety concerns identified.
Sponsor: Neurogen Corporation (Industry)
Responsible Party: Ken Sprenger, MD, MBBCh, Vice President, Clinical Development and Operations, Neurogen Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aplindore-250
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): aplindore 0.05 mg MR total daily dose
  Interventions: Drug: aplindore MR tablets or Placebo
- 2 (Experimental): aplindore 0.1 mg MR total daily dose
  Interventions: Drug: aplindore MR tablets or Placebo
- 3 (Experimental): aplindore 0.25 mg MR total daily dose (to include short titration)
  Interventions: Drug: aplindore MR tablets or Placebo
- 4 (Experimental): aplindore 0.5 mg MR total daily dose (to include short titration)
  Interventions: Drug: aplindore MR tablets or Placebo
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: aplindore MR tablets or Placebo

INTERVENTIONS:
Drug: aplindore MR tablets or Placebo — aplindore MR tablets administered QD for about 4 weeks

SUMMARY:
This is a clinical trial to be conducted at multiple sites in the USA. Patients diagnosed with moderate to severe Restless Legs Syndrome will be randomly allocated to one of 5 treatment arms in the study. The 5 arms include 4 arms with different doses of aplindore MR tablets and 1 placebo arm. The treatment will be taken once a day. The study is blinded and neither patients, nor the investigators, will know what treatment the patient is receiving. Patients will be assigned a dose and will be maintained at that dose for several weeks (2 treatment arms include a short titration period). The entire study will take about 6 weeks. The study will measure how effective aplindore is in decreasing symptoms of Restless Legs Syndrome, and will also assess the safety and tolerability of aplindore.

DETAILED DESCRIPTION:
Two hundred and thirty patients will be randomly assigned to one of five treatment arms in this outpatient study. Of the four aplindore arms, two arms will be titrated over a brief period until the targeted dose is achieved, and then as with the other arms, will be maintained for several weeks. Dosing will take place over a total of about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-85 years;
* Must have a score of ≥20 on the IRLS at Day 1 (Baseline) Visit;
* Have a history of moderate to severe RLS symptoms that disrupted sleep for at least 3 nights per week over at least a 3 month period either immediately before screening or prior to starting any RLS treatment;
* Patients must be off dopamine agonists or any other medications they are taking for RLS for a minimum of one week or 5 half lives of the RLS medication whichever is longer, prior to the Day 1 (Baseline) Visit;
* Patients must be in good general health as determined by a thorough medical history and physical examination (including vital signs), and 12-lead electrocardiogram (ECG);
* Patients must have clinical laboratory values within normal reference range or must not be clinically significantly abnormal as judged by the Investigator at screening;
* Females of childbearing potential must be using an acceptable method of contraception, have a negative serum pregnancy test at screening, and a negative urine pregnancy test at baseline. Acceptable methods of contraception include oral, intrauterine, implantable, injectable contraceptives, hormonal patch, double barrier methods or condoms impregnated with spermicide. After screening, patients using oral contraceptive methods of contraception must agree to add an additional method until 30 days following the last dose of study medication. Women on oral contraceptives must have been using them for at least one month prior to screening;
* Male patients with partners of childbearing potential must agree to use adequate contraception (use of a condom and a spermicidal) during the study and for 3 months after the study;
* Female patients who have been surgically sterilized are eligible if they have a negative pregnancy test at screening and at Baseline;
* If receiving hormone replacement therapy, patients must be on a stable regimen for minimum of 3 months prior to screening;
* Patients must be able to read, understand, and provide written/dated informed consent before enrolling in the study, and must be willing to comply with all study procedures.

Exclusion Criteria:

* Clinically significant unstable medical illness;
* Clinically significant allergic, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease;
* History of non-basal cell cancer or squamous cell cancers or carcinoma in situ of the cervix within 2 years before the screening visit are excluded; for all other cancer diagnoses, patients with a history within 5 years before the screening visit are excluded;
* Patients with plasma ferritin levels less than 10 ng/mL at screening;
* A supine blood pressure > 140/90 mm/Hg at screening or baseline;
* Patients taking OTC or prescription medications that can, in the judgment of the investigator, exacerbate or are the cause of their RLS symptoms will be excluded from the study;
* Patients taking prescription drug therapy or over the counter (OTC) medication for chronic medical conditions other then RLS who are not on stable doses for at least two months prior to screening; patients who are not off any investigational drug for at least 30 days prior to screening;
* History of chronic use of dopamine antagonists for more than 6 months within the past 2 years;
* History or presence of chronic pain other than that associated with RLS. Patients should be excluded if the preponderance of the patient's complaints is related to pain and not associated with the urge to move;
* Clinically significant narcolepsy, parasomnia as an adult, significant circadian rhythm disorder, or secondary causes of RLS, (e.g., uremia or neuropathy);
* Any condition that may affect oral drug absorption;
* Travel across more than three time zones, have an expected change in sleep schedules of 6 hours or more, or have involvement in night shift work within seven days prior to screening through to study completion;
* Any clinically significant abnormal finding at the Screening Visit on physical examination, vital signs, or ECG, as determined by the Investigator; (The QTcF interval must be ≤ 450 msec for males and ≤ 470 msec for females);
* History of allergies, or known sensitivity, hypersensitivity, or adverse reaction to aplindore or structurally similar compounds such as flesinomax, ropinirole or ziprasadone;
* Pregnant or lactating females;
* Recent history (≤ one year) of alcohol or drug abuse, or current evidence of substance dependence or abuse as defined by DSM-IV criteria;
* Regular consumption of large amounts of xanthine-containing substances (i.e. more than 10 cups of coffee or equivalent amounts of xanthine-containing substances per day);
* Prior exposure to aplindore;
* Patients deemed to be in the high risk category for sleep apnea as determined by the Modified Berlin Questionnaire;
* Patients who failed prior treatment with dopamine agonists as evidenced by lack of efficacy at the maximum tolerated dose;
* Patients who test positive at Screening for hepatitis B surface antigen or hepatitis C antiboby or has a history of a positive result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The change from baseline (Day 1) to final (Day 28) on the International Restless Legs Scale (IRLS). | Day 1, Day 14, and Day 28

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - HOPE Research Institute, Phoenix, Arizona
  - Genova Clinical Research, Tuscon, Arizona
  - Excell Research, Inc., Oceanside, California
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Gaylord Sleep Medicine, Wallingford, Connecticut
  - Tampa Bay Medical Research, Clearwater, Florida
  - University Clinical Research Deland, LLC, DeLand, Florida
  - MD Clinical, Hallandale, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Sleep & Behavior Medicine Institute, Vernon Hills, Illinois
  - Community Research & Sleep Management Institute, Crestview Hills, Kentucky
  - Quest Research Institute, Bingham Farms, Michigan
  - Sleep Medicine and Research Center - St Luke's Hospital, Chesterfield, Missouri
  - Wake Research Associates, Raleigh, North Carolina
  - Comunity Reasearch, Cincinnati, Ohio
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Sleep Medicine Associates of Texas, P.A., Dallas, Texas
  - Paragon Research Center, San Antonio, Texas